CLINICAL TRIAL: NCT00606372
Title: Aortocoronary Bypasses in High-Risk Patients (EuroSCORE 6+) With or Without Use of the Cardio-Pulmonary Bypass.
Brief Title: On-Pump vs. Off-Pump CABG in High-Risk Patients (EuroSCORE 6+)
Acronym: PRAGUE 6+
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Charles University, Czech Republic (Other)
Responsible Party: Prof. MUDr. Zbynek Straka, CSc., Kralovske Vinohrady University Hospital
Other Study IDs: 240376
Record Dates: First submitted 2008-01-22; First posted 2008-02-04 (Estimated); Last update posted 2008-02-04 (Estimated); Status verified 2008-01

CONDITIONS: Ischemic Heart Disease; Post-Operative Complications
Keywords: Off-pump; OPCAB; EuroSCORE; high-risk patients; Quality of life; Validity of EuroSCORE
MeSH Terms: conditions — Myocardial Ischemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- 1: Patients with ischemic heart disease, with EuroSCORE 6 additive points and more, operated with use of the cardio-pulmonary bypass
- 2: Patients with ischemic heart disease, with EuroSCORE 6 additive points and more, operated without use of the cardio-pulmonary bypass
  Interventions: Procedure: OPCAB - the off-pump coronary artery bypass

INTERVENTIONS:
Procedure: OPCAB - the off-pump coronary artery bypass — surgical myocardial revascularisation without use of cardio-pulmonary bypass, using stabilising devices on beating heart
  Groups: 2

SUMMARY:
Previous studies comparing on-pump and off-pump operating strategy did only partially demonstrate benefits of the off-pump myocardial revascularisation.In primary end-points (MI, death, renal failure, and so on) there was no significant difference, but in secondary end-points we observed benefits resulting for patients. We would like to show the benefit of the method without extracorporeal circulation in patients with higher and hight operation risk, coming from EuroSCORE classification system (6 points and more).

ELIGIBILITY:
Inclusion Criteria:

* stable form of ischemic heart disease
* unstable angina pectoris
* acute myocardial infarction
* additive EuroSCORE 6 and more
* informed approval of the patient

Exclusion Criteria:

* significant heart valve disease, requesting surgery
* aortic aneurysm requesting surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: People indicated for surgical myocardial revascularisation with high surgical risk
Sampling Method: Probability Sample
Enrollment: 220 (Estimated)
Dates: Start 2006-06; Primary Completion 2008-12 (Actual); Study Completion 2009-12 (Estimated)

PRIMARY OUTCOMES:
death, heart stroke, brain stroke, renal failure, early reoperation | 30 days
heart stroke, brain stroke, death, renal failure, early reoperation | 30 days and 365 days

SECONDARY OUTCOMES:
length of in-hospital stay, blood losses, number of blood-transfusion, new appeared atrial fibrillation, 1-year mortality, quality of life-angina classified by CCS in 1-year follow up, length of mechanical ventilation | 30 days and 365 days

CONTACTS AND LOCATIONS:
Overall Officials: Zbynek Straka, 1, Principal Investigator — Charles University, Prague
Locations (2):
- Czechia (2):
  - Kralovske Vinohrady University Hospital, Prague
  - 2nd Surgical Dpt. of 1st Faculty of Medicine of Charles University, Prague, Prague